CLINICAL TRIAL: NCT04484727
Title: "Lung Barometric Measurements in Normal And in Respiratory Distressed Lungs"
Acronym: LUNAR
Status: Recruiting | Type: Observational
Sponsor: Göteborg University (Other)
Collaborators: Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ALF-75130-5027
Record Dates: First submitted 2020-07-15; First posted 2020-07-24 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Ventilator-Induced Lung Injury; Ventilatory Failure; Ventilator Lung; Ventilation Therapy; Complications; Ventilator Associated Pneumonia
MeSH Terms: conditions — Ventilator-Induced Lung Injury; Hypoventilation; Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ICU-patients in ventilator treatment: Directly after intubation and start of mechanical ventilation, a two-PEEP-step up and down procedure with steps of 5-7 cmH2O each is performed and data on airway pressure and tidal volume changes collected. The data is transferred into a dedicated software for calculation of ΔEELV by cumulative difference in expiratory tidal volume before and during PEEP inflation. Consequently, the lung P/V curve from baseline clinical PEEP to end-inspiration of the highest PEEP level. The PEEP level where clinically used tidal volume has the lowest transpulmonary driving pressure is calculated.
  A one-PEEP-step procedure with a step of 5-7 cmH2O is performed when clinical events such as disconnection of the breathing circuit, posture changes, suctioning, inhalation, CO2 insufflation etc. is performed, and repeated during the whole period of ventilator treatment.
  Interventions: Other: PEEP-step method
- Surgery-patients during general anaesthesia: Directly after intubation and start of mechanical ventilation, a two-PEEP-step up and down procedure with steps of 5-7 cmH2O each, is performed in the same way as described for ICU patients. Data of airway pressure and volumes are transferred into a dedicated software for calculation of ΔEELV by cumulative difference in expiratory tidal volume before and during PEEP inflation. Consequently, the lung P/V curve from baseline clinical PEEP to end-inspiration of the highest PEEP level. The PEEP level where clinically used tidal volume has the lowest transpulmonary driving pressure is calculated.
  A one-PEEP-step procedure with a step of 5-7 cmH2O is performed when clinical events such as disconnection of the breathing circuit, posture changes or suctioning is performed, and before and after implementation of pneumoperitoneum.
  Interventions: Other: PEEP-step method

INTERVENTIONS:
Other: PEEP-step method — By changing PEEP in one or two steps up and down, transpulmonary pressure and the lung P/V curve can be determined using a dedicated software collecting data on tidal-volume changes and pressure changes during the PEEP-changes from the standard monitoring equipment or ventilator.

SUMMARY:
Little is known about how lung mechanics are affected during the very early phase after starting mechanical ventilation. Since the conventional method of measuring esophageal pressure is complicated, hard to interpret and expensive, there are no studies on lung mechanics on intensive care patients directly after intubation, during the first hours of ventilator treatment and forward until the ventilator treatment is withdrawn. Published studies have collected data using the standard methods from day 1 to 3 of ventilator treatment for respiratory system mechanics, i.e. the combined mechanics of lung and chest wall. Consequently, information on lung mechanical properties during the first critical hours of ventilator treatment is missing and individualization of ventilator care done on the basis of respiratory system mechanics, which are not representative of lung mechanics on an individual patient basis. We have developed a PEEP-step method based on a change of PEEP up and down in one or two steps, where the change in end-expiratory lung volume ΔEELV) is determined and lung compliance calculated as ΔEELV divided by ΔPEEP (CL = ΔEELV/ΔPEEP). This simple non-invasive method for separating lung and chest wall mechanics provides an opportunity to enhance the knowledge of lung compliance and the transpulmonary pressure. After the two-PEEP-step procedure, the PEEP level where transpulmonary driving pressure is lowest can be calculated for any chosen tidal volume.

The aim of the present study in the ICU is to survey lung mechanics from start of mechanical ventilation until extubation and to determine PEEP level with lowest (least injurious) transpulmonary driving pressure during ventilator treatment. The aim of the study during anesthesia in the OR, is to survey lung mechanics in lung healthy and identify patients with lung conditions before anesthesia, which may have an increased risk of postoperative complications.

DETAILED DESCRIPTION:
Background:

Acute lung failure requiring respiratory treatment is the most common cause of intensive care in Sweden and the condition has a high mortality rate; approximately 40%. To a large extent, the high mortality rate is due to the patient's underlying disease, e.g. sepsis or trauma but the respiratory treatment itself can also cause mechanical damage to the lungs with the risk of secondary development of acute lung failure and failure in other organ systems such as the liver, kidneys, heart and brain.

In order to reduce the risk and damage of ventilator treatment, it is necessary to improve monitoring of lung function and to develop and evaluate methods for more gentle respiratory treatment.

The studies aim to map the elastic properties of the lungs (pulmonary elastance and transpulmonary drive pressure) in different patient groups, lung healthy and patients with acute lung failure, using the non-invasive PEEP step method. Since the method is non-invasive and is based only on a change in the end expiratory pressure in the ventilator, it can be easily applied during clinical conditions, thus allowing a significant improvement in monitoring and setting of ventilator therapy in both patients under general anesthesia in "major surgery" and patients with acute pulmonary failure in intensive care units.

During general anesthesia, patients lung elasticity will be measured immediately after starting the anesthesia and during surgery and before emergence. In intensive care, the measurement procedure will be applied immediately after the patient has been placed on a ventilator and then during respiratory care when normal intensive care measures take place, such as changing the ventilator setting in terms of breath volume, respiratory rate, end expiratory pressure (PEEP) and similar measures, as well as respiratory suction and inhalations to identify elastic properties within the range normally present in intensive care patients.

Aim:

The aim of the studies is to be able to evaluate lung function during intensive care with new noninvasive measurement methods such as measuring transpulmonary pressure and calculating lung drive pressure, to evaluate lung function during intensive care in order to try to find optimal methods for gentle but effective ventilation of critically ill patients. Studies have previously shown that more gentle respiratory treatment can reduce mortality in respiratory-treated intensive care patients. The development and adaptation of new methods for respiratory treatment and monitoring, can offer better decision support when adjusting airway pressure and volumes, which may ultimately lead to improvements in the form of shorter respiratory time and reduced mortality in respiratory patients. An additional aim is to map normal values of the elastance of the lung ("stiffness") on a population of normal lungs in lung-healthy patients who are sedated for planned surgery.

Main issues:

1. Is the measurement with the PEEP step up and down procedure sufficient to accurately present the lung pressure/volume curve and the transpulmonary drive pressure in respiratory-treated patient populations in surgery and ICU?
2. Is it possible to collect data on a normal population of lung-healthy patients who are sedated for operative surgery as well as in intensive care patients with different degrees of lung failure with the intention of mapping pulmonary elastance/transpulmonary drive pressure and changes in these parameters at initiation of and during respiratory treatment?

Methods:

The PEEP-step method for determining lung elastane: The elastic properties of the lung are measured by increasing PEEP from the clinical baseline level and then lowering the measurement procedure by setting the breath volume to correspond to the lung volume increase that occurs during the PEEP increase. PEEP and tidal volume changes are very common routine measures in both general anesthesia and intensive care. So far, all analysis has been done through manual calculations off-line, but now the measurement procedure and calculations must be automated as far as possible and the transpulmonal drive pressure is presented breath by breath in order to be used for the individualization of the ventilator treatment bedside. This automation is performed in the form of software development. This work is ongoing and expected to be completed in August 2020. Then the PEEP-step method can be implemented and tested in the clinic.

During ten years, in two doctoral theses and four validation studies and additional lung model studies, the investigators have developed an alternative method for measuring the transpulmonary drive pressure, which does not require oesophageal pressure measurement, but only to make a change in the end expiratory pressure (PEEP) in the ventilator and determine the resulting lung volume increase (DEELV) using the ventilator's volume measurement. The elastic properties of the lung (lung elastane, EL) are calculated as DPEEP/DEELV and then the transpulmonary drive pressure is calculated as the volume of breath of the lung elastance, EL x VT. The above additional measurement methods have been evaluated during the last 15 years. Measurement methods collects data from standard monitoring equipment used in clinical anesthesiological practice since the 1980s.

Protocol:

The study is a longitudinal observational study. Measurements will be performed before, during and after respiratory treatment in patients in intensive care units and in surgical units. The measurements take place during the respiratory care period with focus on variations in lung mechanics before and after the procedures included in the clinical routine regarding respiratory settings and other care. Noninvasive measurement methods will be used (see above) of which no one has a negative impact on the patient. Physiological data will be collected from blood gas analyses and monitoring equipment. The monitoring equipment will be connected to a laptop with software that collects continuous clinical data for analysis.

Informed consent: 1) Adult patients who are about to undergo surgery will be consulted at the preoperative assessment approximately 1-2 weeks before surgery about their participation. 2) In adult intensive care patients treated with respiratory therapy, surrogate consent will be prompted. Since it is not previously predicted which patients will be treated on a ventilator in the intensive care unit, the patient's relatives will be asked for informed consent.

For key-references, se References

ELIGIBILITY:
Inclusion Criteria:

* Patients above18 years
* ASA 1-3
* Planned/acute ventilator treatment in ICU or OR

Exclusion Criteria:

* Patients under 18 years
* ASA 4 and above
* severe COPD/emphysema/heart failure
* PEEP>16 and/or FiO2 >80%
* elevated intracranial pressure
* defect coagulation
* non-treated known or suspected pneumothorax

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU-patients or patients in surgery recieving invasive mechancial ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Lung-elastance, changes | Through study completion, an average of 1 year
  Data-collection after intubation, during interventions such as suction, inhalation, posture changes

SECONDARY OUTCOMES:
Hours/Days of ventilator treatment | Through study completion, an average of 1 year
  Registration of Hours/Days of ventilator treatment
Postoperative complications, ICU-complications | Through study completion, an average of 1 year
  Registration of the most common postoperative and ICU-complications

CONTACTS AND LOCATIONS:
Overall Officials: Bengt Nellgård, Prof, Study Chair — Sahlgrenska Academy
Locations (1):
- Sophie Lindgren, Gothenburg, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lundin S, Grivans C, Stenqvist O. Transpulmonary pressure and lung elastance can be estimated by a PEEP-step manoeuvre. Acta Anaesthesiol Scand. 2015 Feb;59(2):185-96. doi: 10.1111/aas.12442. Epub 2014 Dec 2. PMID 25443094
- [Background] Stenqvist O, Grivans C, Andersson B, Lundin S. Lung elastance and transpulmonary pressure can be determined without using oesophageal pressure measurements. Acta Anaesthesiol Scand. 2012 Jul;56(6):738-47. doi: 10.1111/j.1399-6576.2012.02696.x. Epub 2012 Apr 23. PMID 22524531
- [Background] Persson P, Lundin S, Stenqvist O. Transpulmonary and pleural pressure in a respiratory system model with an elastic recoiling lung and an expanding chest wall. Intensive Care Med Exp. 2016 Dec;4(1):26. doi: 10.1186/s40635-016-0103-4. Epub 2016 Sep 20. PMID 27645151
- [Background] Persson P, Stenqvist O, Lundin S. Evaluation of lung and chest wall mechanics during anaesthesia using the PEEP-step method. Br J Anaesth. 2018 Apr;120(4):860-867. doi: 10.1016/j.bja.2017.11.076. Epub 2017 Dec 1. PMID 29576127
- [Background] Stenqvist O, Persson P, Stahl CA, Lundin S. Monitoring transpulmonary pressure during anaesthesia using the PEEP-step method. Br J Anaesth. 2018 Dec;121(6):1373-1375. doi: 10.1016/j.bja.2018.08.018. Epub 2018 Oct 9. No abstract available. PMID 30442269
- [Background] Stenqvist O, Persson P, Lundin S. Can we estimate transpulmonary pressure without an esophageal balloon?-yes. Ann Transl Med. 2018 Oct;6(19):392. doi: 10.21037/atm.2018.06.05. PMID 30460266
- See also: Grivans C., Transpulmonary pressure during mechanical ventilation. Doctoral thesis. ISBN 978-91-628-8832-9. — http://hdl.handle.net/2077/34396
- See also: Persson P. Lung and chest wall properties during mechanical ventilation. Doctoral thesis. ISBN 978-91-7833-224-3 — http://hdl.handle.net/2077/56893